CLINICAL TRIAL: NCT03686085
Title: Effects of Prophylactic Vaginal Dinoprostone Administration Prior to a T380A Intrauterine Device Insertion in Nulliparous Women.
Brief Title: Vaginal Dinoprostone Administration Prior to a T380A Intrauterine Device Insertion in Nulliparous Women.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Samy aly ashour, lecturer in obstetrics and gynecology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: vaginal dinoprostone nullipara
Record Dates: First submitted 2018-09-25; First posted 2018-09-26 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Intrauterine Device
MeSH Terms: interventions — Dinoprostone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dinoprostone arm (Experimental): 1 vaginal tablet of dinoprostone (3mg) (prostin® E2, Pharmacia & Upjohn, Puurs, Belgium) inserted by the study nurse 6 hours before IUD insertion.
  Interventions: Drug: Dinoprostone 3 mg
- placebo (Placebo Comparator): one tablet of placebo inserted by the study nurse 6 hours before IUD insertion.
  Interventions: Drug: placebo vaginal tablet

INTERVENTIONS:
Drug: Dinoprostone 3 mg — 1 vaginal tablet of dinoprostone (3mg) (prostin® E2, Pharmacia & Upjohn, Puurs, Belgium) inserted by the study nurse 6 hours before IUD insertion.
  Arms: dinoprostone arm
Drug: placebo vaginal tablet — 1 vaginal tablet of placebo inserted by the study nurse 6 hours before IUD insertion.
  Arms: placebo

SUMMARY:
To investigate whether vaginal dinoprostone administered before intrauterine device (IUD) insertion reduces failed insertions, insertion-related complications and pain in nulliparous women.

DETAILED DESCRIPTION:
Women may experience pain and technical difﬁculties may be encountered when insertion of an intrauterine device (IUD) is attempted through a narrow cervical canal.IUD insertion- related complications and side effects are more common among women who had never delivered vaginally.n American College of Obstetricians and Gynecologists committee opinion encourages providers to use IUDs as a ﬁrst line of contraception in nulliparous women.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous women aged over 18 years of age requesting a copper IUD for contraception, had a negative pregnancy test.

Exclusion Criteria:

* • a prior pregnancy greater than 20 weeks of duration

  * currently pregnant or were pregnant within 6 weeks of study entry
  * had a prior attempted or successful IUD insertion
  * had a history of a cervical procedure such as cone biopsy, Loop electrosurgical excision procedure, or cryotherapy
  * any World Health Organization Medical Eligibility Criteria category 3 or 4 precaution to an IUD
  * active vaginitis or cervicitis
  * undiagnosed abnormal uterine bleeding
  * pelvic inﬂammatory disease within the last 3 months
  * ﬁbroids or other uterine abnormalities distorting the uterine cavity
  * contraindication to dinoprostone.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2018-09-30 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-10 (Actual)

PRIMARY OUTCOMES:
Provider ease of insertion | 5 minutes
  Provider ease of insertion was evaluated using a visual analog scale from 0 to 10 cm where 0 denotes very easy insertion and 10 denotes a very difficult insertion.

SECONDARY OUTCOMES:
the difference in the pain intensity scores between the study groups | 5 minutes
  the difference in the pain intensity scores between the study groups at IUD insertion BY10 cm visual analog scale score where 0 denotes no pain and 10 denotes the most imaginable pain
insertion time | 10 minutes
  IUD insertion time from speculum in to speculum out

CONTACTS AND LOCATIONS:
Overall Officials: AHMED SAMY, MD, Principal Investigator — Cairo University
Locations (1):
- Faculty of Medicine Cairo University, Giza, Egypt